CLINICAL TRIAL: NCT06193499
Title: A Study on the Effect of High-concentrated Platelet Rich Plasma (PRP) on Osteoarthritis in the Thumb Base.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Maria Wilcke, Associate profesoor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP2.0
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis Thumb
Keywords: CMC-1 joint; thumb basal joint; PRP; Platelet-rich plasma

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: blind fold on participants. No infomration about given treatment to outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet rich plasma (PRP) (Active Comparator): High-concentration PRP injection PRP injection (0,6-1ml). Arthrex ACPmax system.
  Interventions: Procedure: Platelet rich plasma (PRP)
- Placebo (Placebo Comparator): intraarticular saline injection (0,6-1ml)
  Interventions: Other: Placebo

INTERVENTIONS:
Procedure: Platelet rich plasma (PRP) — Intra-articular injection of platelet rich plasma (PRP)
  Arms: Platelet rich plasma (PRP)
Other: Placebo — Intra-articular Saline injection (0,6-1ml)
  Arms: Placebo

SUMMARY:
This is a randomized double-blinded randomized comparison between injection of platelet rich plasma (PRP) and placebo for thumb basale osteoarthritis.

DETAILED DESCRIPTION:
The aim of this study is to evaluate if high-concentration PRP injection decreases pain and disability in patients with thumb base osteoarthritis in the short-term and compare the effect to placebo.90 patients will be inlcuded (45+45). The primary outcome is pain on load (numerical rating scale) after 6 months. Patient-rated outcome measures, pinch grip and key pinch, range of motion of the CMC.1 joint will be assessed before treatment and at 3, 6 and months after the injection. Participants and assessors will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis in the thumb base
* Radiological Eaton Littler class 1-3.
* Clinical signs of thumb base osteoarthritis )pain at palpation of the CMC-1 joint and pain during provocation/grinding test).

Exclusion Criteria:

* Rheumatoid arthritis
* Ongoing infection in the hand or wrist
* History of gout or pseudogout in the hand
* Inability to co-operate with the follow-up protocol (language difficulties, severe psychiatric disorder, cognitive impairment, drug addiction).
* Chronic pain syndrome / centralized pain.
* Intra-articular injection in the affected joint within 6 months.
* Eaton Littler class 4 (symptomatic STT joint osteoarthritis).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain on load in thumb | 6 months after the first injection.
  Pain on load (numerical rating scale (NRS) 0-100, higher score represents more pain)

SECONDARY OUTCOMES:
Patient-rated Wrist and Hand (PRWHE) score | 3 months
  0-100, higher score represents more disability
Patient-rated Wrist and Hand (PRWHE) score | 6 months
  0-100, higher score represents more disability
Patient-rated Wrist and Hand (PRWHE) score | 12 months
  0-100, higher score represents more disability
Nelson thumb score | 3 months
  0-100, lower score represents more symptoms
Nelson thumb score | 6 months
  0-100, lower score represents more symptoms
Nelson thumb score | 12 months
  0-100, lower score represents more symptoms
HAKIR symptom score (HQ-8) | 3 months
  0-100, lower score represents more symptoms
HAKIR symptom score (HQ-8) | 6 months
  0-100, lower score represents more symptoms
HAKIR symptom score (HQ-8) | 12 months
  0-100, lower score represents more symptoms
key pinch and pinch strength | 3 months
  key pinch and pinch strength (kg)
key pinch and pinch strength | 6 months
  key pinch and pinch strength (kg)
key pinch and pinch strength | 12 months
  key pinch and pinch strength (kg)
Radial and palmar abduction | 3 months
  Radial and palmar abduction of the first metacarpal (degrees)
Radial and palmar abduction | 6 months
  Radial and palmar abduction of the first metacarpal (degrees)
Radial and palmar abduction | 12 months
  Radial and palmar abduction of the first metacarpal (degrees)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hand Surgery Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Kieseritzky J, Wilcke M. High-concentrated platelet-rich plasma (PRP) versus placebo in osteoarthritis in the thumb base: study protocol for an assessor-blinded randomized controlled trial. Trials. 2024 Nov 26;25(1):797. doi: 10.1186/s13063-024-08636-2. PMID 39587622